CLINICAL TRIAL: NCT05795270
Title: Multicenter Study on the Role of Neurodegeneration Biomarkers in Characterizing the Severity of Disease and Response to Therapeutic Treatment of Patients With Obstructive Sleep Apnea Syndrome With Residual Excessive Daytime Sleepiness.
Brief Title: Multicenter Study on the Role of Neurodegeneration Biomarkers in Obstructive Sleep Apnea Syndrome With Residual Excessive Daytime Sleepiness.
Acronym: EDS in OSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C121
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Sleep Apnea Syndromes
Keywords: Hypersomnia; Excessive daytime sleepiness; Neurodegeneration biomarkers
MeSH Terms: conditions — Sleep Apnea Syndromes; Disorders of Excessive Somnolence | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleep apnea syndrome with excessive daytime sleepiness
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — Nocturnal ventilotherapy, positional therapy and oro-mandibular devices

SUMMARY:
Excessive daytime sleepiness which still remains after an effective treatment with nocturnal ventilotherapy or with other specific treatments (positional therapy, oro-mandibular devices) in patients with obstructive sleep apnea syndrome has a prevalence of 55% of treated cases, representing a notable theme of clinical and research interest.

In recent years there have been several studies on the use of wakefulness-promoting drugs generally prescribed in patients with narcolepsy, in this disorder with promising results. Right in consideration of the forthcoming approval of these drugs, it is important to find biomarkers able to predict which patients will develop daytime sleepiness resistant to ventilatory treatment. Several studies have highlighted the association between obstructive sleep apnea syndrome and the increase of cerebral amyloid beta deposits, concluding that apnoic disorder can be considered a risk factor for the development of cognitive impairment and Alzheimer';s disease.

In this scenario, it would be useful to identify biological markers able to underline which clinical phenotypes of sleep apnea syndrome are more associated with residual excessive daytime sleepiness and/or cognitive impairment. In recent years several kits for the assay of biomarkers of neurodegeneration have been developed not only in CSF, but also in human serum. Among them, the most important are light chain neurofilaments (NFL), amyloid isoforms 40 and 42 (Ab40 and Ab42). Other biomarkers found in neurodegenerative diseases associated with excessive daytime sleepiness are orexin A (OXA) and histamine (HA).

In this view, the aim of this study is to evaluate the role of biomarkers of neurodegeneration in characterizing disease severity and response to treatment of obstructive sleep apnea syndrome with residual excessive daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Mild or moderate-severe obstructive sleep apnea
* Written informed consent

Exclusion Criteria:

* Other sleep disorders
* Pregnancy or breastfeeding
* Cerebral diseases or neuropsychiatric deficits
* Psychiatric disorders
* Impossibility to provide informed consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sleep apnea syndrome with excessive daytime sleepiness
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-08-24 (Estimated); Study Completion 2023-08-24 (Estimated)

PRIMARY OUTCOMES:
Change in level of light chain neurofilaments | At baseline and after 3 months of treatment
  Plasma level of light chain neurofilaments (NFL)
Change in level of amyloid isoforms 40 and 42 | At baseline and after 3 months of treatment
  Plasma level of amyloid isoforms 40 and 42 (Ab40 and Ab42)
Change in level of daytime sleepiness - Epworth Sleepiness scale | At baseline and after 3 months of treatment
  Level daytime sleepiness - Epworth Sleepiness scale - Minimum 0, Maximum 24

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Oggebbio, Italy